CLINICAL TRIAL: NCT03068507
Title: The Impact of Trimodal Prehabilitation Strategy on Perioperative Functional Capability and Prognosis of Patients Undergoing Thoracoscopic Lobectomy for Lung Cancer：a Randomized Controlled Trail
Brief Title: The Impact of Trimodal Prehabilitation Strategy on Patients Undergoing Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Chairman of anesthesisology department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUMCH8888
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Perioperative; Recovery; Prehabilitation; Thoracoschisis; Lung Cancer; Lobectomy
Keywords: Perioperative; functional capability; Prehabilitation; thoracoscopic lobectomy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: patients were randomly assigned to the prehabilitation group and control group by computer-based random numbers concealed in sealed envelopes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant didn't know their group allocation. The doctor of assessment was blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Trimodal prehabilitation management
  Interventions: Behavioral: Trimodal prehabilitation management
- Control group (No Intervention): The patients will receive the conventional clinical guidance according to Peking Union Medical College Hospital, including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence.

INTERVENTIONS:
Behavioral: Trimodal prehabilitation management — Trimodal prehabilitation strategy includes physical exercise (moderate aerobic exercise combined with resistance exercise and respiratory training ), nutritional suggestion and optimization（whey protein supplement）, and psychological therapy, as well as conventional guidance (including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence).
  Arms: Prehabilitation group

SUMMARY:
The process of enhancing an individual's functional capacity to optimize physiologic reserves before an operation to withstand the stress of surgery has been coined prehabilitation. This is a prospective randomized controlled trail, designed to explore if the patients who take thoracoscopic lobectomy for lung cancer will benefit from family trimodal prehabilitation strategy. Trimodal prehabilitation includes exercise, nutrition supplement and physiology management preoperatively. It starts from the day that patients decide to take the surgery until the day before surgery, lasting 2~3 week in our hospital. And we follow-up patients until 8 weeks after surgery to investigate if trimodal prehabilitation strategy can improve the postoperative functional recovery，reduce complications and improve prognosis.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trail, which focus on the impact of family prehabilitaiton strategy on the patients undertaking thoracoscopic lobectomy for lung cancer.

The process of enhancing an individual's functional capacity to optimize physiologic reserves before an operation to withstand the stress of surgery has been coined prehabilitation. It has been confirm that trimodal prehabilitation strategy including exercise, diet and psychology guidance could improve postoperative functional recovery after surgery for patients undergoing colorectal resection. But there has been no research about the impact of trimodal prehabilitation in other operations.

Although many clinical studies have confirmed that preoperative exercise for patients undergoing lung cancer surgery is safe and useful, but so far there are few studies investigated perioperative functional capability in population undergoing thoracoscopic lobectomy. And no study extends preoperative exercise to trimodal prehabilitation adding nutritional and psychological management. In addition, the prehabilitation strategy in previous studies usually takes 4~8 weeks. However, patient suspected of malignant tumor often wouldn't wait for such a long period. We therefore designed this study to investigate if a 2~3 week family trimodal prehabilitation strategy benefits the patients undergoing thoracoscopic lobectomy for lung caner.

There will be 100 patients awaiting elective thoracoscopic lobectomy for primary lung cancer recruited in this research at Peking Union Medical College Hospital. After informed consent was obtained, the patients will be divided into two groups randomly, the prehibilitation group and control group.

The prehabilitation group will receive an individual trimodal prehabilitation strategy after a complete assessment, including physical exercise, nutritional optimization, and psychological therapy, as well as conventional guidance. The length of prehabilitation was determined by the waiting time till surgery alone. The control group will receive the conventional guidance, including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence. Both of the groups are also provided some useful information about anesthesia and surgery process.

The functional capability will be examined for both groups at several time points (baseline, the day before surgery, 1st, 2nd and 3rd day postoperatively, 4 weeks postoperatively and 8 weeks postoperatively) The primary end point is functional walking capacity as measured by the 6 minutes walking distance (6MWD) 4 weeks postoperatively. The secondary end points include lung function improvement (baseline vs. preoperative) ， self-reported physical activity, health-related quality of life scales and prognosis information (postoperative complications, length of hospital stay, ICU stay time, hospitalization expenses, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient of thoracic surgery department in Peking Union Medical College Hospital
2. From 18 y/o to 70 y/o
3. Suspected of lung cancer
4. Decide to take the elective thoracoscopic surgery in Peking Union Medical College Hospital

Exclusion Criteria:

1. Refuse or fail to cooperate the study (due to any reason)
2. ASA grade ≥ III
3. Unable to tolerate prehabilitaion strategy (including exercise guide, whey protein and psycho-relaxation exercise)
4. Other severe cardio-pulmonary diseases that would affect the 6MWD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
6-minute-walking-distance (6MWD) | 4 weeks postoperatively
  Use 6-minute-walking-distance (6MWD) to evaluate the physical functional capability objectively.

SECONDARY OUTCOMES:
Quality of Life Scale | the 1st, 2nd and 3rd day postoperatively
  Evaluate the intermediate phase of recovery
the version 2 of 12-items Short Form Health Survey(SF 12-v2 | 4 weeks postoperatively
  Evaluate the late phase physical and mental capability recovery after surgery
WHO disability assessment schedule 2.0 (WHODAS 2.0 | 4 weeks postoperatively
  Evaluate the global disability in the late phase of recovery
Hospital Anxiety and Depression Scale (HADS) | 4 weeks postoperatively
  Evaluate the late phase mental capability recovery after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang HUANG, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu Z, Qiu T, Pei L, Zhang Y, Xu L, Cui Y, Liang N, Li S, Chen W, Huang Y. Two-Week Multimodal Prehabilitation Program Improves Perioperative Functional Capability in Patients Undergoing Thoracoscopic Lobectomy for Lung Cancer: A Randomized Controlled Trial. Anesth Analg. 2020 Sep;131(3):840-849. doi: 10.1213/ANE.0000000000004342. PMID 31348053